CLINICAL TRIAL: NCT00565669
Title: Evaluation of Blink Tears and Systane Concomitant With Restasis for the Treatment of Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SEI-07-003
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Dry Eye Syndrome
Keywords: Treatment; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blink Tears (Experimental)
  Interventions: Drug: Cyclosporin A Restasis®; Drug: Blink tears
- Systane (Experimental)
  Interventions: Drug: Cyclosporin A Restasis®; Drug: Systane

INTERVENTIONS:
Drug: Cyclosporin A Restasis®
Drug: Blink tears — blink tears to be used twice a day
  Arms: Blink Tears
Drug: Systane — systane to be used twice a day
  Arms: Systane

SUMMARY:
The purpose of this study is to evaluate the efficacy of Blink Tears and Systane used concomitantly with topical cyclosporine for the treatment of dry eye.

DETAILED DESCRIPTION:
Dry eye is a chronic condition that is believed to afflict more than 3 million patients in the United States.1 Symptoms of dry eye are very bothersome and impact quality of life, reduce work capacity, and may result in poorer psychological health. Also, symptoms of dry eye are associated with a decreased ability to perform activities that require visual attention such as reading and driving a car.2 Patients with dry eye complain most frequently of a scratchy or sandy (foreign body) sensation. Other common symptoms are itching, excessive mucus secretion, inability to produce tears, a burning sensation, photosensitivity, redness, pain, and difficulty in moving the lids. In most patients, the most remarkable feature of the eye examination is the grossly normal appearance of the eye.3 Chronic dry eye disease is associated with an inflammatory mechanism mediated by activated T-cell lymphocytes3 which affects the ocular surface and lacrimal gland.4 The damage caused by dry eye disease may be irreversible, and despite the availability of various tear substitutes, many patients with dry eye syndrome experience corneal injuries with a subsequent reduction in vision.5 Cyclosporin A (Restasis®, Allergan, Irvine, CA) has been shown to significantly reduce the number of activated T-lymphocytes within the conjunctiva6, thereby minimizing the inflammation causing dry eye. Topical cyclosporin A 0.05% ophthalmic emulsion (Restasis®, Allergan, Irvine, CA) increases tear production and improves the quality of naturally produced tears and is the first approved therapeutic agent for the treatment of chronic dry eye and the only treatment modality that addresses the underlying pathology.

In addition to topical therapy with cyclosporine, some patients continue to use artificial tears for occasional relief of residual symptoms. The choice of concomitant tear is important but little research has been published differentiating between the efficacy of these solutions when used concomitantly with topical cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have dry eye.
2. Age: 18 years and older.
3. Males or females
4. Up to grade 3 conjunctival staining.
5. Score of no more than 4 on the Subjective Evaluation of Symptoms of Dryness (SESOD) at screening.
6. Currently using Restasis to treat dry eye syndrome (at least for 3 months prior to enrollment).
7. Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

1. Prior unsuccessful use of topical cyclosporine (defined as patients taking it at least 3 months without improvement.
2. Known contraindications to any study medication or ingredients.
3. Planned use of contact lenses (unless discontinued use more than 30 days prior to randomization.
4. Contact lens use during the active treatment portion of the trial.
5. Active ocular allergies.
6. Ocular surgery within the past 3 months.
7. Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
8. Active ocular diseases or uncontrolled systemic disease (blepharitis patients that are actively being treated or disease that is uncontrollable.
9. Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
10. Participation in (or current participation) any investigational drug or device trial.
11. Conjuctival staining grade 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Medical University of South Carolina, Storm Eye Institute
Locations (1):
- Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blink Tears | Systane
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blink Tears | Systane | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.7) | 67.4 (7.82) | 66.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Schirmer's Scores
Description: The Schirmer score is a score on a scale - minimum is 0 and the highest is 35 mm. Above 15 mm is normal and less than 5 is severe dry eyes. A positive score means there was an improvement, 0 will be no change from baseline and a negative one that there was a decreased in tears. This change was calculated by subtracting the baseline value from the 3 months value (3 mo Schirmer's - baseline Schirmer's = amount of change).
Time Frame: baseline to 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Blink Tears | Systane
Number analyzed (Participants) | 11 | 9
score on a scale | -.30 (2.82) | -1.06 (4.17)

ADVERSE EVENTS:
Arm/Group | Blink Years | Systane
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No